CLINICAL TRIAL: NCT01199757
Title: A Comparison of Patients on AVAMYS ® Versus NASONEX (A Trade Mark of Schering Corporation) and FLIXONASE ® on Key Health Outcome Measures
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Adelphi Real World (Industry)
Responsible Party: Sponsor
Other Study IDs: 114812
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: ocular symptoms; nasal symptoms; Allergic Rhinitis; Symptom Free Days; Quality of Life
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic | interventions — fluticasone furoate; Mometasone Furoate; Fluticasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- FF: Cohort of patients receiving fluticasome furoate
  Interventions: Drug: Fluticasone furoate
- MF: cohort of patients on mometasone furoate
  Interventions: Drug: mometasone furoate
- FP: cohort of patients receiving fluticasone propionate
  Interventions: Drug: fluticasone propionate

INTERVENTIONS:
Drug: Fluticasone furoate — cohort of patients receiving fluticasone furate
  Other Names: AVAMYS™
  Groups: FF
Drug: mometasone furoate — cohort receiving mometasone furoate
  Other Names: NASONEX™
  Groups: MF
Drug: fluticasone propionate — cohort of patients on fluticasone propionate
  Other Names: FLIXONASE™
  Groups: FP

SUMMARY:
Previous publications have indicated that Allergic Rhinitis (AR) patients suffering from both ocular and nasal symptoms have a greater burden of illness and lower quality of life than patients suffering from nasal symptoms alone. Fluticasone furoate (FF) acts against both nasal and ocular symptoms. The purpose of this study was to evaluate the differences in symptom control (both perceptually and objectively) and resource use for patients with current seasonal AR.

DETAILED DESCRIPTION:
* Allergic rhinitis (AR) is a common inflammatory condition of the upper respiratory tract, nasal cavity and eyes affecting up to 20% of the population in the United States and Europe. The bothersome nature of AR symptoms can severely affect daily activities including ability to work and examination performance and impact on quality of life (QoL) and psychosocial well being.
* This study assesses the impact of Fluticasone furoate (FF) on the QoL of seasonal allergic rhinitis (SAR) patients, including the number of symptom-free days (SFD) and quality of life over the last 4 weeks, and compares this with other inhaled nasal steroids (INS): mometasone furate (MF) and fluticasone proprionate (FP).
* Selected physicians provide information including a range of demographic, symptom and treatment details for a number of their SAR patients. The patient themselves are then invited to provide details about their SAR including symptoms, the impact of AR upon their lifestyles, attitudes to treatment and completion of Health Related Quality of Life (HRQoL) instruments.

ELIGIBILITY:
Patient Inclusion Criteria:

* Current Seasonal Allergic Rhinitis sufferer (based on physician judgement)
* Currently receiving prescribed INS treatment (no other treatment restrictions apply)
* Have consumed at least one full prescription on the specified INS treatment
* No comorbid Asthma or COPD diagnosis
* Informed Consent

Exclusion Criteria:

* None specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inclusion criteria for physicians:
  * Qualified after 1965
  * See 3 or more AR patients per week
  * Personally responsible for treatment decisions for patients with AR
  * Gave consent to participate to complete all tasks for the study duration
    90 Primary Care Physicians and 45 allergists, each prospectively recruit 4 consecutive patients with SAR who provided consent to participate, for a total of 540 patients. Each physician completed a patient record form for 2 patients on fluticasone furate, 1 patient on mometasone furate and 1 patient on fluticasone propionate.
Sampling Method: Probability Sample
Enrollment: 540 (Actual)
Dates: Start 2009-07-10 (Actual); Primary Completion 2009-08-01 (Actual); Study Completion 2009-08-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the differences in Symtom Free Days (SFD) in patients receiving FF, MF or FP | 4 weeks

SECONDARY OUTCOMES:
Evaluate the differences in Quality of Life (mini-Rhinoconjunctivitis Quality of Life Questionnaire) in patients receiving FF, MF or FP | 4 weeks
Evaluate the differences in the number of AR treatments used by patients receiving FF, MF or FP | 4 weeks
Evaluate the differences in the number of non-prescribed treatments used by patients receiving FF, MF or FP | 4 weeks
Evaluate the differences in the cost of non-prescribed treatments used by patients receiving FF, MF or FP | 4 weeks
Evaluate the differences in the Pittsburgh Sleep Quality Index in patients receiving FF, MF or FP | 4 weeks
Evaluate the differences in productivitiy (Work Productivity and Activity Impairment Questionnaire) of patients receiving FF, MF or FP | 4 weeks
Evaluate the differences in number of work day lost by patients receiving FF, MF or FP | 4 weeks
Evaluate the differences in the number of physician visits (as reported by patient and doctor) by patients receiving FF, MF or FP | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Higgins V, Kay S, Small M. Physician and patient survey of allergic rhinitis: methodology. Allergy. 2007;62 Suppl 85:6-8. doi: 10.1111/j.1398-9995.2007.01547.x. PMID 17927672
- [Result] Gueron B; Demoly P; Piercy J; Small M. A comparison of patients on Avamys vs Nasonex and Flixonase for Quality of Life and Symptoms Free Days in 3 European countries [Poster 380]. Presented at: XXIXth Congress of the European Academy of Allergy and Clinical Immunology, June 2010, London
- [Derived] Small M, Piercy J, Demoly P, Marsden H. Burden of illness and quality of life in patients being treated for seasonal allergic rhinitis: a cohort survey. Clin Transl Allergy. 2013 Oct 9;3(1):33. doi: 10.1186/2045-7022-3-33. PMID 24107462